CLINICAL TRIAL: NCT00907231
Title: Evaluation of Serial Troponin and Cardiac Multimarkers at the Point of Care in the Emergency Department
Acronym: ESTIMATE
Status: Withdrawn | Type: Observational
Why Stopped: Business Decision
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Director of Clinical Operations, Biosite, Inc
Other Study IDs: BSTE-0112
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Acute Myocardial Infarction; Chest Pain; Acute Coronary Syndrome
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center study to assess the diagnostic accuracy of the Troponin I assay in the Biosite Triage Cardio3 Panel at the point-of-care (POC) in adults presenting to the emergency department with possible acute myocardial infarction (AMI).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of enrollment
* Presenting to the ED within 6 hours from onset of chest discomfort (pain, pressure, tightness, etc) consistent with a possible diagnosis of AMI or ACS and with an initial ECG non-diagnostic for injury (or injury equivalent resulting in emergent reperfusion therapy). (NOTE: Subjects who have chest discomfort that is episodic or stuttering in nature may be included if the ED presentation is within 6 hours of symptom onset.)
* Experiencing at least 30 minutes of chest pain or other anginal equivalent symptoms. (Note: Subjects who have symptoms of shorter duration due to pharmacologic intervention may be included.)

Exclusion Criteria:

* Patient (or Legal Representative) unable or unwilling to provide written informed consent.
* Patient unwilling or unlikely to comply with study procedures, including protocol-specified blood sampling or telephone follow-up at 30 days and 6 months.
* Vulnerable populations as deemed inappropriate for study by site principal investigator.
* ST-elevation or other ECG criteria that result that is diagnostic for AMI and results in patient being sent for percutaneous coronary interventions (PCI) or being treated with thrombolytics6.
* Pulmonary Edema requiring CPAP, BIPAP, or mechanical ventilation
* Tachyarrhythmias (SVT, V-Tach, rapid atrial fib)
* End Stage Renal Disease on Hemodialysis
* Cardiac Arrest prior to arrival
* Implantable Defibrillator firing prior to arrival
* Hemodynamically unstable patients
* Trauma injury to the chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 400 adults presenting to the ED with possible AMI will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Estimated); Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Loyola University Medical Center, Maywood, Illinois
  - Stony Brook University Medical Center, Stony Brook, New York
  - Oregon Health and Sciences University, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Mountain States Health Alliance, Johnson City, Tennessee